CLINICAL TRIAL: NCT03607565
Title: The Association Between a New Parameter Derived From DSA and Outcomes in Cerebral Ischemia
Brief Title: A New Parameter Derived From DSA to Evaluate Cerebral Perfusion
Status: Recruiting | Type: Observational
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Hnn
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- good perfusion in DSA: We introduced a new parameter derived from DSA to evaluate the perfusion in cerebral ischemia.(good perfusion)
- middle perfusion in DSA: We introduced a new parameter derived from DSA to evaluate the perfusion in cerebral ischemia.(middle perfusion)
- poor perfusion in DSA: We introduced a new parameter derived from DSA to evaluate the perfusion in cerebral ischemia.(poor perfusion)

SUMMARY:
This observational study focus on a new parameter of cerebral perfusion derived form digital substraction angiography.

DETAILED DESCRIPTION:
Ischemic cerebrovascular disease is an important cause of death and disability in the world. Digital Subtraction Angiography (DSA) is the golden index for evaluating cerebral blood vessels. We introduced a new parameter derived from DSA to evaluate the perfusion to predict the outcomes in acute stroke with large vessel occlusion.

To study the possible relationship between the new parameter of cerebral perfusion derived from DSA and outcomes in cerebral ischemia（modified Rankin Scale）, we intend to retrospectively analyze the images derived from patients who undergone the DSA and follow-up outcomes（modified Rankin Scale）.

ELIGIBILITY:
Inclusion Criteria:

1. Cerebral ischemia
2. patients undergone DSA

Exclusion Criteria:

1.cerebral hemorrhage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study population is from primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2038-07-15 (Estimated)

PRIMARY OUTCOMES:
the outcomes between good perfusions and poor perfusions | 3 months to 2 years
  Results are reported as odds ratios (ORs) with 95% confidence intervals (CIs).

SECONDARY OUTCOMES:
the outcomes between good perfusions and middle perfusions | 3 months to 2 years
  Results are reported as odds ratios (ORs) with 95% confidence intervals (CIs).

CONTACTS AND LOCATIONS:
Overall Officials: Nannan Han, doctor, Study Director — department of neurology Xi'an No3 Hospital
Locations (1):
- Xi'an No.3 Hospital, Xi'an, Shaanxi, China